CLINICAL TRIAL: NCT05618743
Title: Effect of Non Surgical Therapy on Calprotectin and Periostin Levels in Patients With Periodontitis and Cardiovascular Diseases - An Interventional Study
Brief Title: NSPT on Calprotectin and Periostin Levels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Director of Research and Post Graduate Studies, Professor, Department of Periodontics, Meenakshi Ammal Dental College and Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADC/IEC-I/023/2021
Record Dates: First submitted 2022-02-04; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Chronic Periodontitis; Cardiovascular Diseases; Periodontal Inflammation
MeSH Terms: conditions — Chronic Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Three arm clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): Periodontally and systemically healthy participants (Control group)
- Periodontitis without Cardiovascular disease (Experimental): Periodontitis participants without cardiovascular disease
  Interventions: Procedure: Non Surgical Periodontal Therapy
- Periodontitis with cardiovascular disease (Experimental): Periodontitis participants with cardiovascular disease
  Interventions: Procedure: Non Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non Surgical Periodontal Therapy — Scaling and root planing using scalers and periodontal curettes will be done
  Arms: Periodontitis with cardiovascular disease; Periodontitis without Cardiovascular disease

SUMMARY:
Periodontitis is a chronic inflammatory disease is initiated by the oral microbial biofilm where in the response to this infection is mediated by various intracellular signalling pathways leading to the production of numerous bio-molecules. .

Calprotectin is major cytoplasmic protein expressed in majority by neutrophils and as well seen in gingival epithelial cells, activated macrophages and vascular endothelial cells in minor amounts. Calprotectin is regarded as acute phase protein that increases during a variety of inflammatory diseases like periodontitis, cardiovascular disease, diabetes, rheumatoid arthritis and inflammatory bowel disease. Periostin is a marked anti-inflammatory protein belonging to fascilin family which actively contributed to tissue injury, fibrosis, atherosclerosis and inflammatory diseases Hence this study aims to determine the expression of Calprotectin and Periostin as biomarkers and also as putative risk indicators in generalized chronic periodontitis subjects with or without cardiovascular disease before and after non-surgical therapy.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease is initiated by the oral microbial biofilm where in the response to this infection is mediated by various intracellular signalling pathways leading to the production of numerous bio-molecules. The emerging era of molecular analysis has paved the way to quantify and study the disease markers to which plays a vital role in disease progression. This, in turn, has marked the advent of various studies which employ the use of serum, saliva, gingival crevicular fluid, plaque and tissue samples, etc., to study various diseases in the oral cavity and its relation with systemic diseases.

Several epidemiological studies support an association between high levels of inflammatory biomarkers due to periodontal infections and increased risk and progression of cardio vascular disease. Both periodontitis and cardio vascular disease share various biomarkers expressed in common present in saliva, serum and gingival crevicular fluid which correlates the link of periodontitis with cardiovascular disease.

Calprotectin is major cytoplasmic protein expressed in majority by neutrophils and as well seen in gingival epithelial cells, activated macrophages and vascular endothelial cells in minor amounts. Calprotectin is regarded as acute phase protein that increases during a variety of inflammatory diseases like periodontitis, cardiovascular disease, diabetes, rheumatoid arthritis and inflammatory bowel disease. Calprotectin have been detected in GCF and oral tissues where in initial periodontal therapy can reduce the levels of Calprotectin, but their clinical signiﬁcance has never been investigated in patients with chronic periodontitis and cardiovascular disease.

Among the various matricellular proteins expressed in saliva and GCF, Periostin is a marked anti-inflammatory protein belonging to fascilin family which actively contributed to tissue injury, fibrosis, atherosclerosis and inflammatory diseases. Periostin is commonly found in collagen rich tissues thereby it is thought to affect the production of collagen fibrils. The defensive role of Periostin in periodontal tissues and its expression in periodontitis and cardio vascular disease correlating with before and after non-surgical therapy is less studied which on further exploration might be a potent risk assessment tool linking periodontal and cardiovascular diseases.

While there are studies which have demonstrated the expression of Calprotectin and Periostin in gingival crevicular fluid (GCF) of periodontal patients separately, there are no studies which correlate their interrelationship in periodontitis and cardiovascular disease. Hence this study aims to determine the expression of Calprotectin and Periostin as biomarkers and also as putative risk indicators in generalized chronic periodontitis subjects with or without cardiovascular disease before and after non-surgical therapy.

ELIGIBILITY:
Inclusion Criteria:

• Patients willing to participate in the study. Patients within the age group of 30-65 years. Patients should have ≥ 20 remaining natural teeth. For Group I Systemically healthy, Periodontally healthy subjects with Probing pocket depth (PD) less than 4mm, bleeding on probing (BOP) at ≤15% of tooth sites, no periodontal treatment (Scaling and root planing or periodontal surgery) within the previous 6 months and without evident clinical signs of gingival inflammation. .

For Group II Generalized chronic periodontitis subjects with 30% or more sites with clinical attachment loss (CAL) ≥ 2mm, radiographic evidence of alveolar crestal bone loss ≥ 2mm from the cemento-enamel junction along with cardiovascular disease.

For Group III Systemically healthy, Generalized chronic periodontitis subjects with 30% or more sites with clinical attachment loss (CAL) ≥ 2mm, radiographic evidence of alveolar crestal bone loss ≥ 2mm from the cemento-enamel junction.

Exclusion Criteria:

Subjects with systemic conditions such as type I and type II diabetes mellitus, respiratory diseases, renal disease, liver disease, rheumatoid arthritis, allergy, advanced malignancies and HIV infection will be excluded from the present investigation.

For Group III, subjects on drugs such as corticosteroids, antibiotics, within 6 months of investigation will be excluded.

Current smokers and individuals who quit smoking less than 6 months. Patients who have undergone periodontal therapy within the previous 6 months. Pregnant women (pregnancy may alter the oral flora)

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male participants are included belonging to 30-65 years of age
Enrollment: 45 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction in periodontal parameters | Two years
  Reduction in Periodontal Probing Depth (measured in mm)
Reduction in periodontal variables | Two years
  Reduction in Clinical Attachment Level (measured in mm)
Reduction in periodontal criteria | Two years
  Reduction in Plaque Index (measured in numericals)
Reduction in periodontal variables | Two years
  Reduction in Gingival index (mesured in numericals)

CONTACTS AND LOCATIONS:
Overall Officials: Jaideep Mahendra, MDS,PhD, Principal Investigator — Meenakshi Ammal Dental College and Hospitals
Locations (1):
- Jaideep Mahendra, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaner D, Bernimoulin JP, Dietrich T, Kleber BM, Friedmann A. Calprotectin levels in gingival crevicular fluid predict disease activity in patients treated for generalized aggressive periodontitis. J Periodontal Res. 2011 Aug;46(4):417-26. doi: 10.1111/j.1600-0765.2011.01355.x. Epub 2011 Apr 13. PMID 21488873
- [Background] Arslan R, Karsiyaka Hendek M, Kisa U, Olgun E. The effect of non-surgical periodontal treatment on gingival crevicular fluid periostin levels in patients with gingivitis and periodontitis. Oral Dis. 2021 Sep;27(6):1478-1486. doi: 10.1111/odi.13664. Epub 2020 Oct 23. PMID 33012041